CLINICAL TRIAL: NCT01404754
Title: A Phase 1 Placebo-Controlled, Double-Blind Crossover Study to Assess Psychological Effects of MDMA When Administered to Healthy Volunteers
Brief Title: Psychological Effects of Methylenedioxymethamphetamine (MDMA) When Administered to Healthy Volunteers
Acronym: MT-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MT-1
Record Dates: First submitted 2011-07-19; First posted 2011-07-28 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Psychological Effects of Study Drug
Keywords: MDMA; mood; subjective effects; interpersonal closeness
MeSH Terms: interventions — Lactose; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lactose (Inactive Placebo) (Placebo Comparator): Participant receives inactive placebo during day-long experimental session.
  Interventions: Drug: Lactose (inactive placebo)
- 3,4-methylenedioxymethamphetamine (Active Comparator): Participant receives 120 mg midomafetamine HCl possibly followed by 40 mg midomafetamine HCl during a day-long experimental session.
  Interventions: Drug: midomafetamine HCl

INTERVENTIONS:
Drug: Lactose (inactive placebo) — Placebo in an equivalent weight to midomafetamine HCl will be administered in identical appearing capsules during one of two experimental sessions. An equivalent to the initial and supplemental dose will exist.
  Other Names: placebo
  Arms: Lactose (Inactive Placebo)
Drug: midomafetamine HCl — 120 mg midomafetamine HCl will be administered in opaque capsules at the outside of one of two experimental sessions, and upon mutual agreement between the investigator and participant, 40 mg may be administered 1.5 to 2.5 hours later.
  Other Names: midomafetamine; MDMA; 3,4-methylenedioxymethamphetamine; MDMA HCl
  Arms: 3,4-methylenedioxymethamphetamine

SUMMARY:
The goal of this clinical trial is to study MDMA-assisted therapy in healthy volunteers. The main question it aims to answer is:

Do two sessions of MDMA-assisted therapy result in changes in mood, emotional closeness to self and others, and other psychological symptoms?

Researchers will compare MDMA-assisted therapy to placebo with therapy.

Participants will have a non-drug preparatory session prior to each experimental session and an integrative session after each experimental session. Participants who received MDMA will crossover to receive placebo and placebo participants will crossover to receive MDMA.

DETAILED DESCRIPTION:
This study is a Phase 1 study for up to a hundred people, The information gathered during this study may help us better understand the psychological effects produced by MDMA and how those effects can more effectively be used within a therapeutic context, as with people with PTSD. Participants will be healthy volunteers who have completed a program training them in conducting MDMA-assisted psychotherapy. In this randomized, double blind study, subjects will receive placebo and MDMA during two sessions scheduled at least two days apart in a psychotherapy setting. Mood, self-reported interpersonal closeness, psychological symptoms, blood pressure, heart rate and body temperature will be measured, and personality will be measured prior to the first therapy-like session and two months after the second session.

The study will follow a cross-over design, meaning that all participants will receive both MDMA and placebo, with order of session randomly assigned. Study participants will have a preparatory session prior to each experimental session and an integrative session after each session. The researchers will contact them via telephone one and two months after the second experimental session. By comparing changes in mood, feelings of emotional closeness to the self and others and psychological symptoms after placebo and after MDMA, the investigators hope to learn something about the effects of MDMA on mood, subjective experience and the way we think and feel about others.

ELIGIBILITY:
Inclusion Criteria:

* Engaged in a sponsor-supported program for training therapists to perform MDMA-assisted psychotherapy research
* Are at least 21 years old
* Are willing to follow all rules and restrictions related to study participation, including restrictions on medication use for a week prior to experimental sessions and restrictions on food and alcohol consumption on the day prior to each experimental session
* Are willing to remain overnight at the study site
* Agree to have transportation other than driving themselves after the integrative session on the day after each experimental session
* Are willing to be contacted via telephone for all necessary telephone contacts
* If a woman of childbearing potential, must have a negative pregnancy test and agree to use an effective form of birth control
* Are proficient in speaking and reading English
* Agree to have all clinic visit sessions recorded to audio and video

Exclusion Criteria:

* Are pregnant or nursing, or are women of child bearing potential who are not practicing an effective means of birth control
* Weigh less than 48 kg
* Have used "ecstasy" (material represented as containing MDMA) within 6 months of the MDMA session
* Require ongoing therapy with a psychotropic drug
* Meet DSM-V criteria for substance abuse or dependence for any substance
* Unable to give adequate informed consent
* Upon review of past and current drugs/medication must not be on or have taken a medication that is exclusionary
* Upon review of medical or psychiatric history must not have any current or past diagnosis that would be considered a risk to participation in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-04-09 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | Experimental session approximately six hours after drug administration
  Assesses current mood state
Profile of Mood States (POMS) | Day prior to each experimental session
  Assesses current mood state
Profile of Mood States (POMS) | Day after each experimental session
  Assesses current mood state

SECONDARY OUTCOMES:
Interpersonal closeness measure | Day prior to experimental session
  Visual analog scale assessing emotional closeness to self and four other targets
Interpersonal closeness measure | Day of experimental session approximately six hours post-drug administration
  Visual analog scale assessing emotional closeness to self and four other targets
Interpersonal closeness measure | Day after each experimental session
  Visual analog scale assessing emotional closeness to self and four other targets
Brief Symptom Inventory (BSI) | Day prior to each experimental session
  Self-report measure assessing psychiatric symptoms
Brief Symptom Inventory (BSI) | Day of experimental session prior to drug administration
  Self-report measure assessing psychiatric symptoms
Brief Symptom Inventory (BSI) | Day of experimental session approximately five to six hours after drug administration
  Self-report measure assessing psychiatric symptoms
Brief Symptom Inventory (BSI) | Day after each experimental session
  Self-report measure assessing psychiatric symptoms
Columbia Suicide Severity Rating Scale (adapted C-SSRS) | Day prior to each experimental session
  Clinician-administered measure of suicide risk
Neuroticism Extroversion Openness Personality Inventory | At baseline
  Self-report measure of five personality factors; Neuroticism, extroversion, openness to experience, conscientiousness and agreeableness
Neuroticism Extroversion Openness Personality Inventory | Two months after the second experimental session
  Self-report measure of five personality factors; Neuroticism, extroversion, openness to experience, conscientiousness and agreeableness
Columbia Suicide Severity Rating Scale (adapted C-SSRS) | Day after each experimental session
  Clinician-administered measure of suicide risk
Columbia Suicide Severity Rating Scale (adapted C-SSRS) | One month after the second experimental session
  Clinician-administered measure of suicide risk
Columbia Suicide Severity Rating Scale (adapted C-SSRS) | Two months after the second experimental session
  Clinician-administered measure of suicide risk
Columbia Suicide Severity Rating Scale (adapted C-SSRS) | Day six and 12 of telephone contact after second experimental session
  Clinician-administered measure of suicide risk
Columbia Suicide Severity Rating Scale (adapted C-SSRS) | Day of each experimental session prior to drug administration
  Clinician-administered measure of suicide risk
Columbia Suicide Severity Rating Scale (adapted C-SSRS) | Day of each experimental session approximately five to six hours after drug administration
  Clinician-administered measure of suicide risk
Blood pressure (SBP/DBP) | Throughout each experimental session, every 15 minutes for 6 hours, then every 30 minutes for 2 hours
  Periodic assessment of participant blood pressure during both experimental sessions.
Heart rate (pulse) | Throughout each experimental session, every 15 minutes for 6 hours, then every 30 minutes for 2 hours
  Periodic assessment of participant pulse during both experimental sessions.
Body temperature | Approximately every 60 minutes for each experimental session
  Periodic assessment of participant body temperature during both experimental sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Mithoefer, MD, Study Director — Lykos Therapeutics
Locations (3):
- United States (3):
  - Aguazul Bluewater, Inc., Boulder, Colorado
  - Santa Fe MDMA Therapy Training, LLC, Santa Fe, New Mexico
  - Zen Therapeutic Solutions, Mt. Pleasant, South Carolina